CLINICAL TRIAL: NCT03355326
Title: Evaluation of Routine Administration of Glycerin Suppositories to Improve Bowel Function in Patients With Uncomplicated Gastroschisis
Brief Title: Evaluation of Glycerin Suppositories to Improve Bowel Function in Gastroschisis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to sufficiently recruit candidates
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Alan P. Ladd, Professor of Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IU-IRB-1611267731
Record Dates: First submitted 2017-10-24; First posted 2017-11-28 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Gastroschisis
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Glycerin Suppository Group (Experimental)
  Interventions: Drug: Glycerin Suppository
- Non-suppository Group (No Intervention)

INTERVENTIONS:
Drug: Glycerin Suppository — Glycerin suppository is given once daily beginning after conditions described are met and continued until discontinue conditions are met.
  Arms: Glycerin Suppository Group

SUMMARY:
Gastroschisis is a congenital defect of the abdominal wall that leads to evisceration of various amounts of the abdominal organs. The mainstay of therapy is restoring continuity of the abdominal wall, either through primary closure or with a synthetic graft when primary closure is not feasible.

It has been established that bowel function after repair of gastroschisis is impaired due to the aforementioned pathological processes. Previous studies have shown that the time from surgery to attaining full nutrition through enteral means is a predictor for morbidity in this population. Therefore, numerous therapeutic interventions have been proposed to help hasten bowel function and decrease the time to tolerance of total enteral nutrition. A common, but unproven, technique is the use of glycerin suppositories to stimulate bowel function. The concept of glycerin suppositories is that stimulating colonic activity through the use of the suppository will stimulate small intestinal function. The underlying concept is that improved bowel motility and reduced time to full enteral feeds will reduce the morbidity associated with this disease. While the formation/evacuation of stools is most easily monitored, the main purpose of using these suppositories is to hasten tolerance of nutrition through enteral means.

While the practice of using glycerin suppositories is common in neonates, there is no literature or best-practice guidelines advocating for (or against) their use. A single previous prospective study utilizing glycerin suppositories in premature, low birth weight neonates failed to show any benefit in improving time to tolerate full enteral feeds. At this time, this is the only study investigating the use of glycerin suppositories in any neonatal population, and due to the indications (i.e. premature and low birth weight infants without surgical disease), the findings are not applicable to neonates with gastroschisis. To the authors' knowledge, there are no previous studies or current ongoing studies examining this question. Given this lack of information regarding the efficacy of glycerin suppositories, there is a significant variation in practice among practicing surgeons, including timing of initial administration, frequency of use, and indication to discontinue. Indeed the spectrum ranges from some surgeons who never use glycerin suppositories, to some who prescribe them daily for all gastroschisis patients immediately following surgery.

The purpose of this study will be to determine whether routine use of glycerin suppositories improves bowel function as measured by time to full enteral feeds (primary outcome: defined as enteral feed volume >120mL/kg/day with appropriate weight gain (20-30g/day for two consecutive days)) in neonates with uncomplicated gastroschisis after complete reduction of abdominal viscera. Secondary outcomes include time to first bowel movement and incidence/severity of TPN-induced cholestasis in the study groups.

DETAILED DESCRIPTION:
Gastroschisis is a congenital defect of the abdominal wall that leads to evisceration of various amounts of the abdominal organs. The mainstay of therapy is restoring continuity of the abdominal wall, either through primary closure or with a synthetic graft when primary closure is not feasible. Closure of the abdominal cavity is confounded by prenatal loss of abdominal domain coupled by resultant swelling of the abdominal viscera due to prenatal exposure to amniotic fluid. Additionally, some patients with gastroschisis have other concomitant abnormalities of the bowel (termed complicated gastroschisis) that require additional surgical intervention.

It has been established that bowel function after repair of gastroschisis is impaired due to the aforementioned pathological processes. Previous studies have shown that the time from surgery to attaining full nutrition through enteral means is a predictor for morbidity in this population. Therefore, numerous therapeutic interventions have been proposed to help hasten bowel function and decrease the time to tolerance of total enteral nutrition. A common, but unproven, technique is the use of glycerin suppositories to stimulate bowel function. The concept of glycerin suppositories is that stimulating colonic activity through the use of the suppository will stimulate small intestinal function. The underlying concept is that improved bowel motility and reduced time to full enteral feeds will reduce the morbidity associated with this disease. While the formation/evacuation of stools is most easily monitored, the main purpose of using these suppositories is to hasten tolerance of nutrition through enteral means.

While the practice of using glycerin suppositories is common in neonates, there is no literature or best-practice guidelines advocating for (or against) their use. A single previous prospective study utilizing glycerin suppositories in premature, low birth weight neonates failed to show any benefit in improving time to tolerate full enteral feeds. At this time, this is the only study investigating the use of glycerin suppositories in any neonatal population, and due to the indications (i.e. premature and low birth weight infants without surgical disease), the findings are not applicable to neonates with gastroschisis. To the authors' knowledge, there are no previous studies or current ongoing studies examining this question. Given this lack of information regarding the efficacy of glycerin suppositories, there is a significant variation in practice among practicing surgeons, including timing of initial administration, frequency of use, and indication to discontinue. Indeed the spectrum ranges from some surgeons who never use glycerin suppositories, to some who prescribe them daily for all gastroschisis patients immediately following surgery.

The purpose of this study will be to determine whether routine use of glycerin suppositories improves bowel function as measured by time to full enteral feeds (primary outcome: defined as enteral feed volume >120mL/kg/day with appropriate weight gain (20-30g/day for two consecutive days)) in neonates with uncomplicated gastroschisis after complete reduction of abdominal viscera. Secondary outcomes include time to first bowel movement and incidence/severity of TPN-induced cholestasis in the study groups.

Individuals will be followed from the time of consultation by the Pediatric General Surgery service (i.e. at the time of birth) until initial discharge. Neonates undergo abdominal wall closure and reach full nutrition (via either full enteral, total parenteral nutrition, or a combination of both) prior to discharge.

Patients will approached by a study coordinator (Daisy Nunez or Robert Vandewalle) regarding enrollment, which will occur on the day of, or prior to completion of surgical intervention. Randomization into treatment/control arm, utilizing a block technique, will occur after completion of surgical intervention. While the operating surgeon will technically be unaware of the treatment arm of the patient at the time of surgery, neither the medical staff, study participants/families, or study staff be blinded for this study.

After closure of the abdominal wall children will be cared for according to the same standards used in previous/non-trial patients. The only exception is that the control-group patients will not be allowed to be administered glycerin suppositories at anytime and the treatment- group will receive glycerin suppositories (based upon previously established institutional pharmacy dosing protocols) from the first day after abdominal wall closure until they reach full enteral feeds (as defined as 120mL/kg/d with appropriate weight gain) which will be determined by the surgeon of record. Initiation and advancement of enteral feeds will be based upon on protocol developed for this study and agreed upon the study surgeons, who are responsible for nutritional management of these patients (see attached feeding protocol). Signs of feeding intolerance are outline in the attached feeding protocol. Additional metrics will be recorded in the study data sheet (see attached data collection sheet) this information is routinely collected as a part of normal care for patients with gastroschisis but otherwise no additional interventions will be a part of the study protocol. Because the most common morbidities associated with gastroschisis center on infectious complications and those related to prolonged parenteral nutrition, general indicators for these complications (i.e. laboratory and clinical variables) will be recorded as well.

The electronic patient chart will be reviewed on each patient each weekday of the patient's hospital admission (i.e. real time data collection) and the surgery team/study coordinator will contact the attending of record and/or nursing staff for clarification of any missing data. Both study coordinators will review the dataset independently on a weekly basis to help ensure fidelity of the database and data will be backed up on a twice a week basis.

No additional intervention, interaction, or follow up will be completed after the neonate is discharged from their initial admission as part of this study.

Identified barriers to enrollment included timing of delivery/transfer to Riley Hospital for proper enrollment. This will be addressed by the investigators reviewing the general surgery census list on a daily basis to identify patients early and provide time for patient/family consideration for enrollment. Additional enrollment barriers include language barriers which will be addressed with interpreter requests when available and translator phone when live interpreters are not available and/or not feasible.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uncomplicated gastroschisis
* Gestational age >33 weeks at time of delivery
* Weight >1900g at time of delivery
* Transfer of patient to Riley Hospital for Children prior to any abdominal surgery

Exclusion Criteria:

* Neurological Congenital malformations and/or those known to impair intestinal motility
* Additional congenital gastrointestinal abnormalities requiring surgical intervention
* Congenital Cyanotic heart disease
* Surgical Closure of abdominal wall defect with prosthetic material (e.g. prosthetic or bio-prosthetic mesh)

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ladd, M.D., Principal Investigator — Program Director, Department of General Surgery, Divison of Pediatric Surgery
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-suppository Group: Non-Suppository: No suppository is given beginning after conditions described are met and continued until discontinue conditions are met.
Period: Overall Study
Arm/Group | Glycerin Suppository Group | Non-suppository Group
Started | 9 | 7
Completed | 6 | 4
Not Completed | 3 | 3
Not completed — Protocol Violation | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycerin Suppository Group | Non-suppository Group | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 4 | 10
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 5.5 [2.75 to 6.75] | 4.5 [4.0 to 5.25] | 5.0 [4.0 to 6.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10
Birth weight [Median (Inter-Quartile Range); unit: kg] | 2.39 [2.17 to 2.73] | 2.53 [2.37 to 2.79] | 2.49 [2.23 to 2.75]
Prenatal gastroschisis diagnosis [Number; unit: participants] | 5 | 3 | 8
Size of Silo [Median (Inter-Quartile Range); unit: cm] — Population: one patient did not have silo placed
  cm
    number analyzed (Participants) | 5 | 4 | 9
    (all) | 4.0 [4.0 to 5.5] | 4.0 [4.0 to 4.38] | 4.0 [4.0 to 5.5]

OUTCOME MEASURES:

1. Primary Outcome: Time to Full Enteral Feeds
Description: time from study start time to goal full feeds by enteral route (per oral (PO), orogastric (OG), gastrostomy tube (gtube)).
Time Frame: 2 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Glycerin Suppository Group | Non-suppository Group
Number analyzed (Participants) | 6 | 4
days | 18.5 [14.25 to 22.75] | 17.0 [15.25 to 20.0]
Statistical Analysis 1: Comparison: Glycerin Suppository Group vs Non-suppository Group; Test type: Superiority; p = 0.971, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time to First Bowel Movement
Description: time from study start time after closure to first bowel movement
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Glycerin Suppository Group | Non-suppository Group
Number analyzed (Participants) | 6 | 4
days | 2.5 [2.0 to 3.75] | 3.0 [1.75 to 4.75]
Statistical Analysis 1: Comparison: Glycerin Suppository Group vs Non-suppository Group; Test type: Superiority; p = 0.900, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Hospital Length of Stay
Description: time from admission (birth) to hospital discharge
Time Frame: ~3 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Glycerin Suppository Group | Non-suppository Group
Number analyzed (Participants) | 6 | 4
days | 26.5 [22.5 to 35.25] | 23.5 [21.75 to 27.25]
Statistical Analysis 1: Comparison: Glycerin Suppository Group vs Non-suppository Group; Test type: Superiority; p = 0.648, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Days on Total Parenteral Nutrition (TPN)
Description: total time that patient required Total Parenteral Nutrition (TPN) feeds
Time Frame: 2 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Glycerin Suppository Group | Non-suppository Group
Number analyzed (Participants) | 6 | 4
days | 19.0 [16.5 to 23.75] | 20.5 [17.25 to 24.25]
Statistical Analysis 1: Comparison: Glycerin Suppository Group vs Non-suppository Group; Test type: Superiority; p = 0.967, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants With Sequela of Long Term Total Parenteral Nutrition (TPN) Administration
Description: Any complications related to TPN administration, including TPN-induced cholestasis and hyperbilirubinemia
Time Frame: ~3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Glycerin Suppository Group | Non-suppository Group
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0
Statistical Analysis 1: Comparison: Glycerin Suppository Group vs Non-suppository Group; Test type: Superiority; p > 0.999, Fisher Exact

6. Secondary Outcome: Number of Participants With Infectious Complications
Description: Any complications related to infections during the admission after start of study; these include infections such as line infections, wound infections, pneumonia, and urinary tract infection (UTI)
Time Frame: ~3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Glycerin Suppository Group | Non-suppository Group
Number analyzed (Participants) | 6 | 4
Participants | 2 | 2
Statistical Analysis 1: Comparison: Glycerin Suppository Group vs Non-suppository Group; Test type: Superiority; p > 0.999, Fisher Exact

7. Secondary Outcome: Number of Participants With Post-operative Complications
Description: Any complications during the admission after start of study; these include anything including infections, necrotizing enterocolitis (NEC), small bowel obstruction (SBO), and Total Parenteral Nutrition (TPN)-induced cholestasis.
Time Frame: ~3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Glycerin Suppository Group | Non-suppository Group
Number analyzed (Participants) | 6 | 4
Participants | 2 | 2
Statistical Analysis 1: Comparison: Glycerin Suppository Group vs Non-suppository Group; Test type: Superiority; p > 0.999, Fisher Exact

ADVERSE EVENTS:
Time Frame: through study completion, an average [or up to] 3 months.
Arm/Group | Glycerin Suppository Group | Non-suppository Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 2/6 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glycerin Suppository Group (N=6) | Non-suppository Group (N=4)
Postop infection (Infections and infestations) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT03355326/Prot_SAP_002.pdf
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT03355326/ICF_001.pdf